CLINICAL TRIAL: NCT04278560
Title: Modulating Brain Activity to Improve Goal-directed Physical Activity in Older Adult
Brief Title: Modulating Brain Activity to Improve Goal-directed Physical Activity in Older Adults
Acronym: Stim-Fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-2019-26
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Aging
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Behavioral intervention plus tDCS (Experimental): This intervention will consist of a two-month, personalized, goal-based counseling approach to promote physical activity. Over the first two weeks of the behavioral intervention, participants will also received 10, once-daily, 20-minute sessions of transcranial direct current stimulation (tDCS) designed to increase the excitability of the left dorsolateral prefrontal cortex.
  Interventions: Device: Transcranial direct current stimulation (tDCS); Behavioral: Behavioral intervention to increase physical activity
- Behavioral intervention plus sham stimulation (Active Comparator): This intervention will consist of a two-month, personalized, goal-based counseling approach to promote physical activity. Over the first two weeks of the behavioral intervention, participants will also received 10, once-daily, 20-minute sessions of sham stimulation.
  Interventions: Device: Sham stimulation; Behavioral: Behavioral intervention to increase physical activity

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — tDCS will be delivered via six gel electrodes with placement and current parameters optimized based on a standard brain to maximize the average normal component of the generated electric field over the left dlPFC. Current delivered by anyone electrode will never exceed 2.0 mA; the total amount of current from all electrodes will not exceed 4 mA. Each 20-minute session will begin and end with a 60-second ramp up/down of current amplitude to maximize comfort.
  Arms: Behavioral intervention plus tDCS
Device: Sham stimulation — An 'active' sham will be used in which very low-level currents are transferred between the same electrodes used in the active condition throughout the 20-minute session. However, currents will be designed to mimic the cutaneous sensations induced by tDCS yet not significantly influence cortical tissue.
  Arms: Behavioral intervention plus sham stimulation
Behavioral: Behavioral intervention to increase physical activity — Study staff will complete face-to-face and telephone counseling sessions with each participant, tailored to their state of readiness to increase physical activity levels. The participant will be provided with a goal to increase their average daily step count by 20% from baseline. The staff member will review the participant's stated barriers to exercise and provide them with a list of strategies they may use to augment their step counts throughout each day. Bi-weekly face-to-face counseling sessions will then be completed to review and discuss activity performance and answer any questions the participant may have regarding their efforts to increase physical activity.

SUMMARY:
Although the majority of older adults are aware of the compelling evidence that regular exercise is critical to the maintenance of health into old age, most do not meet recommendations for daily exercise. This lack of engagement in 'goal-directed' physical activity stems from numerous interrelated factors including lack of motivation, depressed mood, and cognitive "executive" impairments that diminish one's ability to regulate behavior over time. Intriguingly, each of these factors has been linked to the function of brain networks that include the left dorsolateral prefrontal cortex (dlPFC). Transcranial direct current stimulation (tDCS) is a noninvasive and safe means of modulating the excitability of specific brain regions and their connected neural networks. tDCS designed to facilitate the excitability of the left dlPFC has been shown to improve motivation, mood, and multiple aspects of executive function in healthy adults. The investigators thus hypothesize that tDCS holds promise to increase goal-directed physical activity in older adults. This project aims to conduct a pilot randomized controlled trial on the feasibility and effects of a 2-week, 10-session tDCS intervention targeting the left dlPFC, combined with behavioral intervention aimed at increases daily physical activity, on physical activity over a two-month follow-up period, in relatively sedentary older adults without overt illness or disease.

ELIGIBILITY:
Inclusion Criteria:

* Must live within subsidized housing in the Boston area
* Self-report of exercising, on average, less than 150 minutes of at least moderate-intensity exercise per week, as determined by phone-screen completion of the International Physical Activity Questionnaire-Short Form (IPAQ short)

Exclusion Criteria:

* An inability to ambulate without the assistance of another person (canes or walkers allowed)
* Self-report of physician-diagnosed dementia, more than moderate cognitive impairment defined as a Montreal Cognitive Assessment (MoCA) score <21, or an inability to understand the study protocol as determined by study staff
* A clinical history of stroke, Parkinson's disease or parkinsonian syndromes, multiple sclerosis, normal pressure hydrocephalus or other movement disorder affecting gait
* Any report of severe lower-extremity arthritis or physician-diagnosis of peripheral neuropathy
* Use of antipsychotics, anti-seizure, benzodiazepines, or other neuroactive medications
* Severe depression defined by a Geriatric Depression Scale score greater than 11
* Any report or physician-diagnosis of schizophrenia, bipolar disorder or other psychiatric illness
* Any unstable medical condition
* Resting systolic blood pressure is higher than 180 mmHg
* Contraindications tor tDCS, including reported seizure within the past two years, use of neuro-active drugs, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemaker, etc.), or the presence of any active dermatological condition, such as eczema, on the scalp

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Manor, PhD, Principal Investigator — Hebrew SeniorLife
Locations (1):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The HSL Institute for Aging Research will promote the development of new research and new investigators by making the data available to outside investigators. The database will include longitudinal demographic, clinical, functional, physiologic, and brain imaging data, from all participants.
  All data will be stripped of primary identifiers and entered into a master database. All data collection procedures, variable definitions and codes, field locations, and frequencies will be documented in a separate file.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The investigators will make the data and associated documentation available once summary data are published or otherwise made available, starting six months after publication.
Access Criteria: The investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: 1) a commitment to using data only for research purposes and not to identify any particular participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed. The availability of data will be advertised over the Internet through websites maintained by Hebrew SeniorLife and Harvard Medical School.
  All investigators wishing to access the data will submit a brief proposal describing their research project, data needs, regulatory approvals, and mechanisms to assure patient confidentiality. Upon affirmative review by the Principal Investigator and co-investigators of this study, a data-sharing agreement will be signed and the requesting investigators will be given a working data file and appropriate documentation.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants signed the informed consent at the in-person screening but withdrew prior to the baseline assessment and were never randomized.
Groups:
- Behavioral Intervention Plus tDCS: This intervention will consist of a two-month, personalized, goal-based counseling approach to promote physical activity. Over the first two weeks of the behavioral intervention, participants will also received 10, once-daily, 20-minute sessions of transcranial direct current stimulation (tDCS) designed to increase the excitability of the left dorsolateral prefrontal cortex.
  Transcranial direct current stimulation (tDCS): tDCS will be delivered via six gel electrodes with placement and current parameters optimized based on a standard brain to maximize the average normal component of the generated electric field over the left dlPFC. Current delivered by anyone electrode will never exceed 2.0 mA; the total amount of current from all electrodes will not exceed 4 mA. Each 20-minute session will begin and end with a 60-second ramp up/down of current amplitude to maximize comfort.
  Behavioral intervention to increase physical activity: Study staff will complete face-to-face and telephone counseling sessions with each participant, tailored to their state of readiness to increase physical activity levels. The participant will be provided with a goal to increase their average daily step count by 20% from baseline. Bi-weekly face-to-face counseling sessions will then be completed to review and discuss activity performance and answer any questions the participant may have regarding their efforts to increase physical activity.
Period: Overall Study
Arm/Group | Behavioral Intervention Plus tDCS | Behavioral Intervention Plus Sham Stimulation
Started | 16 | 16
Completed | 15 | 13
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Intervention Plus tDCS | Behavioral Intervention Plus Sham Stimulation | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (7.8) | 81.2 (6.0) | 78.6 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change of Daily Step Counts From Baseline
Description: Absolute change in averaged daily step counts from two-week baseline (first two weeks, week 1-2). The specific periods are 1) absolute change in averaged daily step counts in week 3 and 4 from baseline, 2) absolute change in averaged daily step counts at week 5 and 6, from baseline, 3) absolute change in averaged daily step counts in week 7 and 8 from baseline, and 4) absolute change in averaged daily step counts in week 9 and 10 from baseline.
Time Frame: Week 3-4, Week 5-6, Week 7-8, and Week 9-10.
Measure: Mean (Standard Error); unit: Steps per day
Arm/Group | Behavioral Intervention Plus tDCS | Behavioral Intervention Plus Sham Stimulation
Number analyzed (Participants) | 15 | 13
Steps per day
  Week 3-4 | 842 (281) | 194 (219)
  Week 5-6 | 1099 (405) | 408 (443)
  Week 7-8 | 1299 (439) | 721 (284)
  Week 9-10 | 1476 (519) | 866 (448)
Statistical Analysis 1: Comparison: Behavioral Intervention Plus tDCS vs Behavioral Intervention Plus Sham Stimulation; Test type: Superiority; p = 0.009, ANOVA — Repeated Measures Two-Way ANOVA: Group, Time, Group x Time, and controlled by Baseline Step Counts; Mean Difference (Net) = 385.3

2. Secondary Outcome: Motivation - External Regulation Score
Description: External Regulation Score was calculated from the Exercise Self-Regulation Questionnaire (SQR-E). External regulation refers to motivation based on external sources such as incentives or coercion. Introjected regulation refers to motivation from an internalized, pressuring voice that was not accepting it as one's own. The External Regulation Score ranges from 4 to 28. The higher scores mean a better outcome.
Time Frame: Baseline; Week 4; Week 10
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Behavioral Intervention Plus tDCS | Behavioral Intervention Plus Sham Stimulation
Number analyzed (Participants) | 15 | 13
score on a scale
  Baseline | 5.9 (0.7) | 5.7 (0.7)
  Week 4 | 8.1 (1.5) | 5.3 (0.5)
  Week 10 | 8.1 (1.2) | 5.8 (0.9)
Statistical Analysis 1: Comparison: Behavioral Intervention Plus tDCS vs Behavioral Intervention Plus Sham Stimulation; Test type: Superiority; p = 0.03, ANOVA; We used change from baseline for this analysis. Two-Way Repeated Measure ANOVA: Group, Time, Group x Time, and controlled baseline; Mean Difference (Net) = 1.2

3. Secondary Outcome: Timed Up-and-Go (TUG)
Description: A common field test of mobility
Time Frame: Baseline; Week 4; Week 10
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Behavioral Intervention Plus tDCS | Behavioral Intervention Plus Sham Stimulation
Number analyzed (Participants) | 15 | 13
seconds
  Baseline | 10.9 (0.7) | 12.8 (1.1)
  Week 4 | 11.0 (0.6) | 12.9 (0.9)
  Week 10 | 10.7 (0.7) | 12.4 (0.9)
Statistical Analysis 1: Comparison: Behavioral Intervention Plus tDCS vs Behavioral Intervention Plus Sham Stimulation; Test type: Superiority; p = 0.4, ANOVA; We used change from baseline for the analysis. Two-Way Repeated Measure ANOVA: Group, Time, Group x Time, and controlled baseline; Mean Difference (Net) = 0.19

4. Secondary Outcome: Trail Making Test (TMT) - A
Description: Trail making test (TMT) A is a neuropsychological test of visual attention. The test requires the patient to connect randomly positioned numbered circles in numeric order as quickly as possible. It provides information about visual search speed and speed of processing. The test reliability for TMT A is 0.82. Time is measured in seconds.
Time Frame: Baseline; Week 4; Week 10
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Behavioral Intervention Plus tDCS | Behavioral Intervention Plus Sham Stimulation
Number analyzed (Participants) | 15 | 13
Seconds
  Baseline | 36.3 (4.0) | 39.9 (3.0)
  Week 4 | 29.8 (2.1) | 39.8 (2.8)
  Week 10 | 32.4 (3.6) | 38.4 (2.5)
Statistical Analysis 1: Comparison: Behavioral Intervention Plus tDCS vs Behavioral Intervention Plus Sham Stimulation; Test type: Superiority; p = 0.016, ANOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 3.1

5. Secondary Outcome: Trail Making Test (TMT) - B
Description: Trail Making Test (TMT) - B is a neuropsychological test of task switching. The test requires the participants to connect the circles in numeric and alphabetic order as quickly as possible, alternating between numbers and letters. It provides information about executive function. The test reliability for TMT-B is 0.93. Time is measured in seconds.
Time Frame: Baseline; Week 4; Week 10
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Behavioral Intervention Plus tDCS | Behavioral Intervention Plus Sham Stimulation
Number analyzed (Participants) | 15 | 13
Seconds
  Baseline | 101.6 (13.5) | 106.2 (11.0)
  Week 4 | 101.4 (15.0) | 122.4 (19.9)
  Week 10 | 86.7 (10.4) | 113.0 (19.7)
Statistical Analysis 1: Comparison: Behavioral Intervention Plus tDCS vs Behavioral Intervention Plus Sham Stimulation; Test type: Superiority; p = 0.17, ANOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 9.94

6. Secondary Outcome: Montreal Cognitive Assessment (MoCA) Total Score
Description: Global cognitive function. The range for this test is 0-30, with higher score representing better outcome.
Time Frame: Baseline; Week 4; Week 10
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Behavioral Intervention Plus tDCS | Behavioral Intervention Plus Sham Stimulation
Number analyzed (Participants) | 15 | 13
score on a scale
  Baseline | 25.8 (0.5) | 24.0 (0.5)
  Week 4 | 24.6 (0.7) | 24.4 (0.9)
  Week 10 | 24.8 (0.6) | 24.3 (0.8)
Statistical Analysis 1: Comparison: Behavioral Intervention Plus tDCS vs Behavioral Intervention Plus Sham Stimulation; Test type: Superiority; p = 0.1, ANOVA; [statistical method as in outcome 2, analysis 1]; Median Difference (Net) = 0.6

7. Secondary Outcome: Geriatric Depression Scale (15-item)
Description: Number of depressive symptoms. The range for this test is 0-15, with lower score representing better outcome.
Time Frame: Baseline; Week 4; Week 10
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Behavioral Intervention Plus tDCS | Behavioral Intervention Plus Sham Stimulation
Number analyzed (Participants) | 15 | 13
score on a scale
  Baseline | 2.1 (0.4) | 2.7 (0.6)
  Week 4 | 1.1 (0.4) | 2.1 (0.6)
  Week 10 | 1.4 (0.4) | 1.5 (0.4)
Statistical Analysis 1: Comparison: Behavioral Intervention Plus tDCS vs Behavioral Intervention Plus Sham Stimulation; Test type: Superiority; p = 0.7, ANOVA; [statistical method as in outcome 2, analysis 1]; Median Difference (Net) = 0.07

8. Secondary Outcome: Completion Rate for Brain Stimulation Sessions
Description: Ten stimulation sessions were planned for each participant over two weeks. This outcome presents the percentage of the completed brain stimulation sessions.
Time Frame: Week 4
Measure: Mean (Standard Error); unit: percentage of comleted sessions
Arm/Group | Behavioral Intervention Plus tDCS | Behavioral Intervention Plus Sham Stimulation
Number analyzed (Participants) | 15 | 13
percentage of comleted sessions | 98 (1) | 99 (1)
Statistical Analysis 1: Comparison: Behavioral Intervention Plus tDCS vs Behavioral Intervention Plus Sham Stimulation; Test type: Superiority; p = 0.46, t-test, 2 sided

9. Secondary Outcome: Completion Rate for Behavior Sessions
Description: Four bi-weekly behaviors sessions were planned for each participant over two months. This outcome presents the percentage of the completed behavior sessions.
Time Frame: Week 10
Measure: Mean (Standard Error); unit: percentage of comleted sessions
Arm/Group | Behavioral Intervention Plus tDCS | Behavioral Intervention Plus Sham Stimulation
Number analyzed (Participants) | 15 | 13
percentage of comleted sessions | 97 (2) | 100 (0)
Statistical Analysis 1: Comparison: Behavioral Intervention Plus tDCS vs Behavioral Intervention Plus Sham Stimulation; Test type: Superiority; p = 0.16, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 22 weeks
Arm/Group | Behavioral Intervention Plus tDCS | Behavioral Intervention Plus Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16 | 2/16
Other Adverse Events (participants affected / at risk) | 11/16 | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Intervention Plus tDCS (N=16) | Behavioral Intervention Plus Sham Stimulation (N=16)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Intervention Plus tDCS (N=16) | Behavioral Intervention Plus Sham Stimulation (N=16)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Coronavirus infection (Infections and infestations) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Mole excision (Surgical and medical procedures) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Opthalmic migraine (Nervous system disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bed bug infestation (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Allergy to chemicals (Immune system disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blepharoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT04278560/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT04278560/SAP_002.pdf